CLINICAL TRIAL: NCT05731362
Title: An Early Supported Discharge Model of Care for Older Adults Admitted to Hospital: a Protocol for a Descriptive Cohort Study
Brief Title: An ESD Model of Care for Older Adults Admitted to Hospital: a Protocol for a Descriptive Cohort Study
Status: Withdrawn | Type: Observational
Why Stopped: Change in study design
Sponsor: University of Limerick (Other)
Responsible Party: Sponsor
Other Study IDs: 112/2022
Record Dates: First submitted 2023-01-20; First posted 2023-02-16 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Aging; Hospitalization; Function
Keywords: older adults; early supported discharge; cohort study; hospitalised; patient discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MDCIT Intervention — The MidWest Multidisciplinary Community Intervention Teams (MDCIT) comprise of specialist, healthcare teams that provide a rapid and integrated response to a patient with an acute episode of illness who requires enhanced services/acute intervention for a defined short period of time. This is provided in the patient's home after an acute hospital admission, thereby facilitating early discharge. The MDCIT intervention is composed of occupational therapy, physiotherapy, and healthcare assistants, with nursing support as required.
  The MDCIT therapists aim to make their first visit to patients within 24-48 hours of hospital discharge. Patients receive two-three visits per week, over a period of two to four weeks dependant on the patient's rehabilitation needs. Upon discharge from the MDCIT service, patients can be referred to community services as indicated by therapists.

SUMMARY:
The MidWest multidisciplinary Community Intervention Teams (MD-CIT) comprise of specialist, healthcare teams that provide a rapid and integrated response to a patient with an acute episode of illness who requires enhanced services/acute intervention for a defined short period of time in the MidWest of Ireland. This is provided in the patient's home, thereby facilitating early discharge from the acute hospital setting.

The investigators are performing an evaluation of the MDCIT service provided to older adults admitted to UL Hospitals Group. The investigators will assess patients in hospital, at 30 days and at a six months.

ELIGIBILITY:
Inclusion Criteria:

* Older adults ≥ 65 years who are discharged home (community dwelling) from ULHG with a referral to the MDCIT service between December 2022 and June 2023 will be deemed eligible for recruitment

Exclusion Criteria:

* Those aged < 65 years discharged home from ULHG and referred to the MDCIT service
* Those deemed to not have decision making capacity to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adults admitted to general medical and surgical wards, trauma/orthopaedic wards and acute medical assessment units and subsequently discharged home with MDCIT support will be included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Functional Ability | This will be measured at baseline.
  Function will be measured using the Barthel Index (BI). The BI scores a patient from 0-20, with a higher score indicating greater independence.
Functional Ability | This will be measured at 30 days.
  Function will be measured using the Barthel Index (BI). The BI scores a patient from 0-20, with a higher score indicating greater independence.
Functional Ability | This will be measured at 180 days.
  Function will be measured using the Barthel Index (BI). The BI scores a patient from 0-20, with a higher score indicating greater independence.

SECONDARY OUTCOMES:
Frailty Score | This will be measured at baseline.
  Frailty will be measured using the Clinical Frailty Scale (CFS). The CFS screens for frailty in older adults, with a minimum score of 1 considered least frail and a maximum score of 9 indicating severe frailty.
Frailty Score | This will be measured at 30 days.
  Frailty will be measured using the Clinical Frailty Scale (CFS). The CFS screens for frailty in older adults, with a minimum score of 1 considered least frail and a maximum score of 9 indicating severe frailty.
Frailty Score | This will be measured at 180 days.
  Frailty will be measured using the Clinical Frailty Scale (CFS). The CFS screens for frailty in older adults, with a minimum score of 1 considered least frail and a maximum score of 9 indicating severe frailty.
Patient Quality of Life | This will be measured at baseline.
  Quality of Life will be measured using the EQ-5D-5L. This questionnaire asks a patient to rate their overall perceived health from a scale of 0-100 (0 = very poor; 100 = excellent).
Patient Quality of Life | This will be measured at 30 days.
  Quality of Life will be measured using the EQ-5D-5L. This questionnaire asks a patient to rate their overall perceived health from a scale of 0-100 (0 = very poor; 100 = excellent).
Patient Quality of Life | This will be measured at 180 days.
  Quality of Life will be measured using the EQ-5D-5L. This questionnaire asks a patient to rate their overall perceived health from a scale of 0-100 (0 = very poor; 100 = excellent).
Quality of Care | This will be measured at 30 days.
  Quality of Care will be measured using the Patient Assessment of Integrated Elderly Care. Patients are asked 20 questions across a Likert scale from 'none at all' to 'always.'
Quality of Care | This will be measured at 1800 days.
  Quality of Care will be measured using the Patient Assessment of Integrated Elderly Care. Patients are asked 20 questions across a Likert scale from 'none at all' to 'always.'
Unscheduled ED Attendance(s) | This will be measured at 30 days.
  ED hospital databases will be searched to identify ED attendances.
Unscheduled ED Attendance(s) | This will be measured at 180 days.
  ED software will be searched to identify ED attendances.
Unscheduled Hospital Admission(s) | This will be measured at 30 days.
  ED and hospital software will be searched to identify admissions.
Unscheduled Hospital Admission(s) | This will be measured at 180 days.
  ED and hospital software will be searched to identify admissions.
Nursing Home Admission(s) | This will be measured at 30 days.
  Hospital software will be searched to identify patients admitted to nursing homes.
Nursing Home Admission(s) | This will be measured at 180 days.
  Hospital software will be searched to identify patients admitted to nursing homes.
Mortality | This will be measured at 30 days.
  Hospital software will be searched to identify patients who pass away.
Mortality | This will be measured at 180 days.
  Hospital software will be searched to identify patients who pass away.

CONTACTS AND LOCATIONS:
Overall Officials: Cathryn Ryan, Principal Investigator — MidWest Community Healthcare
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided